CLINICAL TRIAL: NCT00535691
Title: A Randomised, Multi-centre, Double-blind, Pharmacokinetic Study of Tacrolimus Ointment (0.03%) in Paediatric Patients (Aged 3 Months to 24 Months) With Atopic Dermatitis Following First and Repeated Once Daily or Twice Daily Application of the Tacrolimus Ointment
Brief Title: Tacrolimus Ointment Pharmacokinetics in Infants With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FG-506-06-32
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Tacrolimus ointment 0.03% once daily, placebo once daily
  Interventions: Drug: Tacrolimus Ointment 0.03%
- 2 (Active Comparator): Tacrolimus ointment 0.03% twice daily
  Interventions: Drug: Tacrolimus Ointment 0.03%

INTERVENTIONS:
Drug: Tacrolimus Ointment 0.03% — Twice daily, 14 days treatment.
  Other Names: Protopic 0.03%
  Arms: 2
Drug: Tacrolimus Ointment 0.03% — Once daily, 14 days treatment.
  Arms: 1

SUMMARY:
The purpose of this study is to estimate the systemic exposure to tacrolimus in infants with atopic dermatitis after repeated application of tacrolimus ointment. Efficacy of tacrolimus ointment, evaluated by examination of treated areas, will also be measured.

DETAILED DESCRIPTION:
This is a multi-centre, double-blind, randomised phase II pharmacokinetic study in infants (3 - 24 months old) suffering from atopic dermatitis and requiring treatment with mid potency topical steroids. Patients will primarily be stratified into three groups according to percentage body surface area to be treated and subsequently randomised into treatment groups of once a day (UID) or twice a day (BID) tacrolimus ointment (0.03%) regimens. There will ultimately be a total of six groups. The study will be conducted on an out-patient basis, with each patient's parent/legal representative administering the ointment at home. However all medications on days 1 and 14 will be applied in the clinic by the Investigator or his/her designee, as will the morning application on day 4. The ointment application period will be two weeks with a follow-up period of four days. All patients enrolled into the study, who applied at least one dose of study medication and who benefited from treatment will be given the opportunity to enter a long-term study to follow (FG-506-06-33).

The patient will be entered into one of the following three groups:

Stratification Group I Application area of 5 - 20% Stratification Group II Application area of > 20 - 40% Stratification Group III Application area of > 40%

Within these groups the patients will be randomised to either UID or BID.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 3 and 24 months old on Day 1.
* The patient has atopic dermatitis requiring treatment with mid potent topical steroids.
* Patient's disease involves a percentage area to be treated greater than or equal to 5% of the total body surface area

Exclusion Criteria:

* Patient has clinically infected atopic dermatitis.
* Patient has a history of more than two courses of systemic corticosteroid treatment

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2003-04; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Estimate the systemic exposure to tacrolimus after first and repeated application of 0.03% tacrolimus ointment in paediatric patients with atopic dermatitis stratified by application area and randomised to once a day (UID) or twice a day (BID) treatment. | Day 1 and 14

SECONDARY OUTCOMES:
Efficacy of tacrolimus ointment, evaluated by examination of treated areas. | Day 4, 14 and 18

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma GmbH
Locations (8):
- Canada (3):
  - Halifax
  - Vancouver
  - Waterloo
- Helsinki, Finland
- Ireland (2):
  - Drogheda
  - Dublin
- Riga, Latvia
- London, United Kingdom